CLINICAL TRIAL: NCT01480648
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses of BI 144807 Powder in Bottle (1 to 1200 mg) in Healthy Male Volunteers in a Randomised, Single-blind, Placebo-controlled Trial
Brief Title: Single Rising Dose Study of BI 144807 Powder in Bottle in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1313.1; 2011-002560-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (2):
- BI144807 (Experimental): Subjects receive a single oral dose of BI144807solution
  Interventions: Drug: BI 144807
- Placebo (Placebo Comparator): Subjects receive a single oral dose of placebo solution
  Interventions: Drug: BI 144807 Placebo

INTERVENTIONS:
Drug: BI 144807 Placebo — Placebo that represents BI drug
  Arms: Placebo
Drug: BI 144807 — single dose (low to high dose)
  Arms: BI144807

SUMMARY:
This first-in-man trial forms the basis for potential clinical development of BI 144807 in the indications of asthma and allergic rhinitis. The safety, tolerability, pharmacokinetics, and pharmacodynamics of single rising doses of BI 144807 will be assessed in healthy male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
All adverse events | up to 14 days postdose
Number of participants with clinically significant changes in vital signs | up to 14 days postdose
Number of participants with clinically significant changes in ECG | up to 14 days postdose
Number of participants with clinically significant changes in laboratory tests | up to 14 days postdose
Number of participants with clinically significant changes in physical examination | up to 14 days postdose
Number of participants tolerating BI 144807 | up to 14 days postdose

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72h postdose
tmax (time from dosing to maximum measured concentration) | up to 72h postdose
AUC0-8 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72h postdose
AUC(0-tz) (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72h postdose
t1/2 (terminal half-life of the analyte in plasma) | up to 72h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1313.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany